CLINICAL TRIAL: NCT04207970
Title: Evaluating Adapted Structured Clinical Management for People With a Diagnosis of Personality Disorder
Status: Completed | Type: Observational
Sponsor: Camden and Islington NHS Trust (Other Government)
Responsible Party: Principal Investigator, Andrew White, Clinical Psychologist, Camden and Islington NHS Trust
Other Study IDs: 262702
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Personality Disorders
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clients under PDS Community Team: 27 adult clients under PDS Community Team
  Interventions: Other: Adapted Structured Clinical Management

INTERVENTIONS:
Other: Adapted Structured Clinical Management — Adapted form of a previous Evidence Based Treatment- adapted to local context, in light of input from service-users and commissioners.

SUMMARY:
Camden and Islington NHS Foundation Trust in London has a Personality Disorder Service (PDS) which offers a number of evidence-based interventions to people with a diagnosis of Personality Disorder. One team in the PDS, the Community Team, offers an adapted form of Structured Clinical Management (SCM; Bateman and Kravitz, 2013). As these adaptations are novel, this study aims to formally explore the effectiveness of this intervention, through a sample of clients under the team, with outcomes (proxy measures of distress such as inpatient admissions) pre- and post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Allocated to a care coordinator at the PDS for greater than one year (a reasonable time period for therapeutic rapport to form and the effect of the intervention to manifest).

Exclusion Criteria:

* No existing notes for one year prior to allocation.
* No primary diagnosis of Personality Disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of Personality Disorder, under the care of Camden and Islington PDS.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Proxy measures of client distress | One year pre-referral and one year post-allocation
  Inpatient admissions, safeguarding concerns, crisis centre contacts, crisis house admissions, criminal justice contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew White, Principal Investigator — Camden and Islington NHS Trust
Locations (1):
- Camden and Islington Personality Disorder Service, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No